CLINICAL TRIAL: NCT04107727
Title: A 2:1 Randomized Phase II Trial to Compare the Efficacy and Safety of Standard Chemotherapy Plus Quizartinib Versus Standard Chemotherapy Plus Placebo in Adult Patients With Newly Diagnosed FLT3 Wild-type AML
Brief Title: Trial to Compare Efficacy and Safety of Chemotherapy/Quizartinib vs Chemotherapy/Placebo in Adults FMS-like Tyrosine Kinase 3 (FLT3) Wild-type Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Dynamic Science S.L. (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QUIWI
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Quizartinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib; Cytarabine; Idarubicin

STUDY DESIGN:
Intervention Model Description: Safety run-in phase: multicenter, prospective, open-label.
  Phase II: multicenter, prospective, randomized, placebo-controlled, double-blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized into 1 of the 2 treatment groups (quizartinib or placebo) in a 2:1 ratio. The randomization will be stratified by age (<60 vs. ≥60 years old) at the time of diagnosis of AML. Neither the subjects nor any of the Investigators, Sponsor, or contract research organizations (CROs) will be aware of the treatments received. An independent biostatistician, not otherwise part of the study team, will generate the randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quizartinib (Experimental): Induction: Cytarabine continuous IV infusion 200 mg/m2 (days 1-7), Idarubicin IV infusion 12 mg/m2 (days 1-3), oral quizartinib (dose defined in safety run-in phase) 14 days (8-21) (dose will be halved with strong CYP3A inhibitor), up to 2 cycles of 35 days.
  Consolidation: Cytarabine IV infusion 1,5-3 g/m2 (days 1, 3, 5), oral quizartinib (dose defined in safety run-in phase) 14 days (6-19) (dose will be halved with strong CYP3A inhibitor), up to 4 cycles of 35 days.
  Maintenance: oral quizartinib 60mg/day (dose will be halved with strong CYP3A inhibitor), up to 12 cycles of 28 days
  Interventions: Drug: Quizartinib; Drug: Cytarabine; Drug: Idarubicin
- Placebo (Placebo Comparator): Induction: Cytarabine continuous IV infusion 200 mg/m2 (days 1-7), Idarubicin IV infusion 12 mg/m2 (days 1-3), oral placebo (dose defined in safety run-in phase) 14 days (8-21) (dose will be halved with strong CYP3A inhibitor), up to 2 cycles of 35 days.
  Consolidation: Cytarabine IV infusion 1,5-3 g/m2 (days 1, 3, 5), oral placebo (dose defined in safety run-in phase) 14 days (6-19) (dose will be halved with strong CYP3A inhibitor), up to 4 cycles of 35 days.
  Maintenance: oral placebo 60mg/day (dose will be halved with strong CYP3A inhibitor), up to 12 cycles of 28 days.
  Interventions: Drug: Placebo oral tablet; Drug: Cytarabine; Drug: Idarubicin

INTERVENTIONS:
Drug: Quizartinib — Induction: oral quizartinib (dose defined in safety run-in phase) 14 days (8-21) (dose will be halved with strong CYP3A inhibitor), up to 2 cycles of 35 days.
  Consolidation: oral quizartinib (dose defined in safety run-in phase) 14 days (6-19) (dose will be halved with strong CYP3A inhibitor), up to 4 cycles of 35 days.
  Maintenance: oral quizartinib 60mg/day (dose will be halved with strong CYP3A inhibitor), up to 12 cycles of 28 days.
  Arms: Quizartinib
Drug: Placebo oral tablet — Induction: oral placebo (dose defined in safety run-in phase) 14 days (8-21) (dose will be halved with strong CYP3A inhibitor), up to 2 cycles of 35 days.
  Consolidation: oral placebo (dose defined in safety run-in phase) 14 days (6-19) (dose will be halved with strong CYP3A inhibitor), up to 4 cycles of 35 days.
  Maintenance: oral placebo 60mg/day (dose will be halved with strong CYP3A inhibitor), up to 12 cycles of 28 days.
  Arms: Placebo
Drug: Cytarabine — Induction: Cytarabine continuous IV infusion, 200 mg/m2 (days 1-7), up to 2 cycles of 35 days.
  Consolidation: Cytarabine IV infusion, 1,5-3 g/m2 (days 1, 3, 5), up to 4 cycles of 35 days.
Drug: Idarubicin — Induction: Idarubicin IV infusion 12 mg/m2 (days 1-3), up to 2 cycles of 35 days.

SUMMARY:
Randomized phase II trial to compare the efficacy and safety of standard chemotherapy plus quizartinib versus standard chemotherapy plus placebo in adult patients with newly diagnosed FLT3 wild-type Acute Myeloid Leukemia

DETAILED DESCRIPTION:
Multicenter, prospective, randomized, placebo-controlled, double-blinded phase II trial to assess the efficacy and safety of an oral quizartinib vs. placebo containing front-line chemotherapy-based schedule in FMS-like tyrosine kinase 3 internal tandem duplications (FLT3-ITD) wild-type Acute Myeloid Leukemia patients.

The trial will be conducted in two phases:

An open-label safety run-in phase: Cytarabine 200 mg/m2 (days 1-7), Idarubicin 12 mg/m2 (days 1-3) Quizartinib 60 mg/d x 14 days (30mg with strong Cytochrome P450 Family 3 Subfamily A (CYP3A) inhibitor) in a total of 9 patients, being observed during 1 cycle of induction to define the final dose for the randomized phase.

A randomized double-blinded phase 2:1 quizartinib (at the established dose) vs. placebo.

Experimental Arm: Cytarabine 200 mg/m2 (days 1-7), Idarubicin 12 mg/m2 (days 1-3) Quizartinib 60 mg/d x 14 days (30mg with strong CYP3A inhibitor) Standard Arm: Cytarabine 200 mg/m2 (days 1-7), Idarubicin 12 mg/m2 (days 1-3) Placebo 60 mg/d x 14 days (30mg with strong CYP3A inhibitor)

272 patients will be included in this phase.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with national, local, and institutional guidelines. The patient must provide informed consent before the first screening procedure. The patient and the investigator must sign informed consent form.
2. Diagnosis of untreated AML (according to the World Health Organization (WHO) 2008/2016 definition)
3. Age ≥ 18 and ≤70 years old at the time of screening
4. Non-FLT3-ITD (allelic ratio <0.03) at diagnosis
5. Considered eligible to receive intensive chemotherapy as per investigator judgment
6. Eastern Cooperative Oncology Group (ECOG) 0-2
7. No contraindications for quizartinib
8. The subject is receiving standard "7+3" induction chemotherapy regimen as specified in the protocol
9. No severe organ function abnormalities
10. Not included in other first-line trials
11. Cardiac ejection fraction ≥ 45% assessed by echocardiography or multiple-gated acquisition (MUGA).
12. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use reliable methods of contraception upon enrollment, during the treatment period and for 3 months following the last dose of investigational drug or cytarabine, whichever is later
13. Male patients must use a reliable method of contraception (if sexually active with a female of child-bearing potential) upon enrollment, during the treatment period, and for 3 months following the last dose of investigational drug or cytarabine, whichever is later
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with a genetic diagnosis of acute promyelocytic leukemia
2. Age <18 years or >70 years
3. ECOG performance status of 3 or 4
4. Prior treatment for AML, except for the following allowances:

   c) Leukapheresis d) Treatment for hyperleukocytosis with hydroxyurea
5. Blastic phase of bcr/abl chronic myeloid leukemia.
6. Presence of an associated active and/or uncontrolled malignancy:

   - Patients with another neoplastic disease, for whom the Investigator has a clinical suspicion of active disease at the time of enrollment. Note: Patients with adequately treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia are eligible for this study. Hormonal or adjuvant therapies will be allowed for breast cancer or prostate cancer as long as they are on a stable dose for at least 2 weeks before the first dose.
7. Known active and not controlled hepatitis B or hepatitis C infection. In the event of a positive viral load, please consult with the Sponsor
8. Known human immunodeficiency virus (HIV) infection (HIV testing is not required as part of this study)
9. Presence of any severe psychiatric disease or physical condition that, according to the physician´s criteria, contraindicates the inclusion of the patient into the clinical trial
10. Serum creatinine ≥ 250 μmol/l (≥ 2.5 mg/dL) (unless it is attributable to AML activity)
11. Bilirubin, alkaline phosphatase, or Serum glutamic oxaloacetic transaminase (SGOT) > 3 times the normal upper limit (unless it is attributable to AML activity)
12. Uncontrolled or significant cardiovascular disease, including any of the following:

    1. Symptomatic bradycardia of fewer than 50 beats per minute, unless the subject has a pacemaker;
    2. QT Comparison of Fridericia's (QTcF) >450 msec at Screening. Note: QTcF will be derived from the mean of triplicate readings;
    3. Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
    4. Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥ 110 mmHg;
    5. History of clinically relevant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes)
    6. History of a second (Mobitz II) or third-degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker)
    7. An ejection fraction <45%
    8. History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening
    9. History of New York Heart Association Class 3 or 4 heart failure
    10. Right bundle branch and left anterior hemiblock (bifascicular block), complete left bundle branch block
13. History of hypersensitivity to any excipients in the quizartinib/placebo tablets
14. Females who are pregnant or breastfeeding
15. Any patients with known significant impairment in gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of quizartinib.
16. Active acute or chronic Graft-Versus-Host-Disease (GVHD) requiring prednisone >10 mg or equivalent corticosteroid daily.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Event-free survival rate | Through study completion, an average of 5 years
  Time from randomization to the date of the occurrence of any of the following events: CR/CRi after 1 or 2 induction cycles, death in CR/CRi or relapse, whichever occurs the first

SECONDARY OUTCOMES:
Maximum dose tolerated (MDT) and recommended phase 2 dose (Safety run-in phase) | At the end of Cycle 1 of Induction and up to 59 days (Safety run-in phase)
  To determine the maximum dose tolerated (MDT) and the recommended phase 2 dose
Composite Complete Remission (CR/CRi) with minimal residual disease (MRD) negativity | Through study completion, an average of 5 years
  The proportion of subjects with complete response or complete remission with incomplete blood count recovery with Minimal residual disease negative
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 5 years
  Adverse events between experimental quizartinib containing schedule and standard arm
Disease-free survival | Through study completion, an average of 5 years
  To compare the time from the first documentation of remission to the documentation of disease recurrence or death.
Overall survival | Through study completion, an average of 5 years
  The number of days from randomization until death from any cause
Cumulative incidence of Relapse | Through study completion, an average of 5 years
  To compare the time from the date of first Complete Response until date of hematological or extramedullary relapse

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, Principal Investigator — Hospital Universitari i Politecnic La Fe
Locations (44):
- Spain (44):
  - Complejo Hospitalario Universitario de A Coruña, Santiago de Compostela, A Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General Univesitario de Castellón, Castellon, Castellón
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Quirón Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario de Galdakao, Galdakao, Vizcaya
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Complejo Hospitalario Lucus Augusti, Lugo
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Regional Universitario Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Universitario de Navarra, Pamplona
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Complejo Hospitalario Regional Virgen del Rocío, Seville
  - Hospital Nuestra Señora del Prado, Talavera de la Reina
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico Universitario Valencia, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
  - Hospital Txagorritxu, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montesinos P, Rodriguez-Veiga R, Bergua JM, Algarra Algarra JL, Botella C, Rodriguez-Arboli E, Bernal T, Tormo M, Calbacho M, Salamero O, Serrano J, Noriega V, Lopez-Lopez JA, Vives S, Lopez-Lorenzo JL, Colorado M, Vidriales MB, Garcia Boyero R, Olave MT, Herrera Puente P, Arce O, Barrios M, Jose Sayas M, Polo M, Gomez-Roncero MI, Barragan E, Ayala R, Chillon C, Calasanz MJ, Paiva B, Boluda B, Casas-Aviles I, Lloret-Madrid P, Sanchez MJ, Rodriguez-Medina C, Cuevas L, Raposo-Puglia JA, Mateos MC, Olivares M, Martinez-Chamorro C, Alonso N, Suarez S, Sanchez-Vadillo I, Sole Rodriguez M, Gonzalez BJ, Martinez-Frances A, Cuello R, Fernandez A, Martinez-Cuadron D, Labrador J; PETHEMA group; PETHEMA Group. Quizartinib for Newly Diagnosed FLT3-Internal Tandem Duplication-Negative AML: The Randomized, Double-Blind, Placebo-Controlled, Phase II QUIWI Study. J Clin Oncol. 2026 Jan;44(1):42-53. doi: 10.1200/JCO-25-01841. Epub 2025 Oct 13. PMID 41082703